31/12/2020

Steba Biotech SA Sponsor:

Study title:

Study of the Efficacy, Safety and Quality of Life after TOOKAD  $^{\circledR}$  Soluble Vascular Targeted Photodynamic therapy (VTP) for Minimally .Invasive Treatment of Localized Intermediate Risk Prostate Cancer

Study number: CLIN1601 PCM204

**SAP version:** 04 January 2021 (Version 1.0)

> DocuSigned by: andrew Vickers

Signer Name: Andrew Vickers

Signing Reason: I approve this document

Signature Date 4-Jan-2021 | 08:30:29 PST 723A6CE189A149B19E542AC8A75D3229

Trial Biostatistician:

Name: Andrew Vickers Function: Biostatistician

Company: Memorial Sloan Kettering Cancer Center

City: New York Country: USA

DocuSigned by:

Simon Hogan

Signer Name: Simon Hogan

Signing Reason: I approve this document Signatyra Date: 04-Jan-2021 | 17:31:54 CET D37CB9E9BA4D47E7A83985580847AB82

Name: Simon Hogan

Function:

Company: Steba Biotech

City: Country:

# Confidentiality statement:

Sponsor's representative:

The information provided in this document is strictly confidential.

The Recipients of the SAP must not disclose the confidential document and any related information to other persons.

In addition, they must keep this confidential document in a controlled environment which prevents unauthorized access to the document.

CLIN1601 PCM204 SAP 

# Statistical Analysis Plan (SAP)

# 31/12/2020

# TABLE OF CONTENTS

| LIST OF ABBREVIATIONS | |
|-----------------------------------------------------------|----|
| ntroduction | |
| Study Objectives, endpoints and Design | |
| Objectives | |
| Primary objective | |
| Secondary objectives | |
| Endpoints | |
| Primary endpoint | |
| Secondary endpoints | |
| Study design | |
| Assessments and study duration | |
| Planned sample size | |
| nterim analyses | |
| Analysis populations | 6 |
| Safety population (Safety) | |
| Efficacy population | |
| Statistical Considerations and analysis | 6 |
| Derived variables | |
| Handling of missing data and/or invalid data and outliers | |
| IEF questionnaire | |
| PSS questionnaire | 8 |
| Statistical plan and methods | 8 |
| Background characteristics | |
| Subject disposition | |
| Demographic and baseline characteristics | |
| Treatment modalities | 8 |
| Efficacy analysis | 8 |
| Primary efficacy analysis | 8 |
| Secondary efficacy analysis | |
| Safety analysisSafety analysis | 9 |
| Adverse events | |
| Clinical laboratory evaluation | |
| /ital signs | |
| Physical exam | |
| Changes from the planned analysis in study protocol | |
| References | 10 |

#### Statistical Analysis Plan (SAP)

31/12/2020

# Explanation

#### LIST OF ABBREVIATIONS

Abbreviation or special term

AE Adverse Event

ATC Anatomical Therapeutic Classification

BMI Body Mass Index
CRF Case Report Form

CTC Common Terminology Criteria

ECG Electrocardiogram

IIEF International Index of Erectile Function
IPSS International Prostate Symptom Score

LDI Light Density Index

MedDRA Medical Dictionary for Regulatory Activities

MRI Magnetic Resonance Imaging
NCI National Cancer Institute

OC Observed Cases
PP Per Protocol

**PSA** Prostate Specific Antigen SAE Serious Adverse Event SAP Statistical Analysis Plan SD Standard Deviation SE Standard Error SOC System Organ Class **TNM Tumor Node Metastasis TRUS** Trans Rectal Ultrasound VAS Visual Analogue Scale

VTP Vascular-Targeted Photodynamic therapy

WHO World Health Organization

CLIN1601 PCM204 SAP 

#### Introduction

The purpose of this statistical analysis plan (SAP) is to provide an analytic framework, which addresses analyses in support of the protocol objectives. This analysis plan is based on the protocol of the PCM204 study as protocol version 6.0 dated 1st October 2018 (MSKCC IRB# 17 070(2)).

# Study Objectives, endpoints and Design

# **Objectives**

# **Primary objective**

The primary objective of the study i sis to evaluate for the absence of biopsydetectable Gleason grade 4 or 5 prostate cancer on 12- month, post-treatment biopsy following TOOKAD® Soluble- VTP in men with Gleason score 7 (3+4) prostate cancer.

# Secondary objectives

The secondary objectives of the study are:

- To describe the rate of responders, with response defined as the absence of any Gleason pattern 4 or 5 biopsy on or before months 24, 36, 48 and 60. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of Gleason pattern 4 or 5, the subject will be considered to have responded
- 2. To describe the rate of responders, with response defined as the absence of any prostate cancer on biopsy on or before months 3, 12, 24, 36, 48 and 60. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of any cancer, the subject will be considered to have responded
- 3. To describe the rate of responders, with response defined as the absence of any Gleason grade 4 or 5 biopsy on or before months 12, 24, 36, 48 and 60 in the treated lobe. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of gleason grade 4 or 5, the subject will be considered to have responded
- 4. To describe the rate of responders, with response defined as the absence of any prostate cancer on biopsy on or before months 3, 12, 24, 36, 48 and 60 in the treated lobe. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of any cancer, the subject will be considered to have responded
- 5. To describe the change in biopsy results between 3, 12, 24, 36, 48 and 60 months after TOOKAD® Soluble-VTP.
- 6. To describe changes in urinary and erectile function and their potential impact on QOL using International Prostate Symptom Score (IPSS) and International Index of Erectile Function (IIEF) questionnaires up to 60 months
- 7. To describe the occurrence of adverse events of TOOKAD® Soluble VTP treatment in patients with localized prostate cancer
- 8. To describe the occurrence of severe prostate cancer-related events: cancer extension to T3, metastasis and prostate cancer-related death

CLIN1601 PCM204 SAP 

- To document the occurrence of secondary prostate cancer therapies following VTP treatment
- 10. To describe changes in PSA from blood samples following TOOKAD® Soluble-VTP.

# **Endpoints**

# **Primary endpoint**

The primary efficacy variable is the result of the Month 12 biopsy, in which success is defined by absence of detectable Gleason grade 4 or 5 prostate cancer.

The primary endpoint will be analysed as a dichotomous outcome, i.e., success (absence of any histology result positive for Gleason 4 or 5 prostate cancer at 12 months) or failure (presence of at least one result positive for Gleason grade 4 or 5 prostate cancer at 12 months).

# Secondary endpoints

- Binary response to treatment defined as the absence of any Gleason grade 4 or 5 biopsy on or before months 24, 36, 48 and 60. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of Gleason grade 4 or 5, the subject will be considered to have responded
- Binary response to treatment defined as the absence of any Gleason grade 4 or 5 biopsy on or before months 12, 24, 36, 48 and 60 in the treated lobe. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of Gleason grade 4 or 5, the subject will be considered to have responded
- Binary response to treatment defined as the absence of any prostate cancer on biopsy on or before months 3, 12, 24, 36, 48 and 60. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of any cancer, the subject will be considered to have responded
- Binary response to treatment defined as the absence of any prostate cancer on biopsy on or before months 3, 12, 24, 36, 48 and 60 in the treated lobe. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of any cancer, the subject will be considered to have responded
- Changes in biopsy result between 3, 12, 24, 36, 48 and 60 months after the procedure
- Patients' reported outcome measures (PROMs) impairment: urinary symptoms using IPSS and erectile functions using IIEF prior to treatment beginning and then 1, 3, 6, 12, 24, 36, 48 and 60 months after completing treatment.

Quality of life is assessed using validated questionnaires. The IPSS comprises seven questions on the urinary symptoms plus one general question about the QOL related to urinary symptoms, whereas the IIEF comprises 15 questions. For both questionnaires, patients self-rate their responses: for the IPSS, using a six-point scale where 0 indicates 'none' or 'normal', whereas 5 indicates the worst response; for the

CLIN1601 PCM204 SAP 

IIEF, using a five- or six-point scale where 0 indicates 'no sexual activity', and 5 indicates the best response (questions 1 to 10), or where 1 indicates the worst response and 5 the best response (questions 11 to 15).

Rate of adverse events following treatment

# Study design

## Assessments and study duration

This is a single center, single-arm, open-label, 60-month follow-up phase IIb clinical trial with assessments at 3, 12, 24, 36, 48 and 60 months.

#### Planned sample size

For an assumed true response rate of 83.6%, we can discount a response rate of 70% at a one-sided alpha of 10%, with a power of 80% if we have a sample size of 44 patients.

# Interim analyses

No interim analysis is planned during the study. However, this does not preclude an analysis of the primary endpoint after all data on this endpoint are available, that is after the last patients have completed the Month 12 visit. No further analysis of the primary endpoint will be done after results of this analysis have been published.

# **Analysis populations**

# Safety population (Safety)

The safety population includes all who received any amount of TOOKAD® Soluble or initiated any study treatment related procedure (including initiation of pre-procedure anesthesia). The safety population will be used for all safety endpoints.

# Efficacy population

The efficacy population will include patients who complied with the protocol for inclusion criteria and exclusion and follow-up received the appropriate dose of TOOKAD® Soluble, LDI and energy delivered and underwent the VTP procedure, receiving the ascribed dose of TOOKAD® Soluble and light, had no major protocol deviations and provided data at the 12 month biopsy. A "major" protocol deviation is defined as one which, in the opinion of the PI, could importantly influence the result of the 12 months biopsy and which is adjudicated before the 12-month biopsy.

## Statistical Considerations and analysis

#### Derived variables

#### Total number of positive cores

The total number of positive cores observed during follow-up is calculated by adding the maximum number of positive cores observed in each of the right and left lobes.

#### Time to stage progression

The time to progression will be calculated from the date of the procedure to the date of stage progression defined as the earliest date of onset of one of the following events, whichever occurs the earliest:

• Extracapsular extension confirmed with tissue sampling

CLIN1601 PCM204 SAP 

- Seminal vesical invasion confirmed with tissue sampling
- Metastasis based on tissue confirmation with biopsy or post-mortem evaluation
- Cancer-related death will be assessed based on tissue confirmation with biopsy or post-mortem evaluation.

Subjects with no documented stage progression will be censored at the date of the last available on study disease assessment

# Time to additional radical therapy (Days)

The time to additional radical therapy will be calculated from the date of treatment to the date of initiation of the first radical therapy. If a subject did not receive any additional radical therapy during the study then the time to additional radical therapy for this subject will be censored at the study termination date.

# Time since diagnosis (Months)

The time since diagnosis will be calculated from the date of diagnosis to the date of treatment.

Age (years) = (date of informed consent – date of birth)/365.25 rounded to the lowest integer.

# **Body Mass Index (BMI)**

BMI  $(kg/m^2)$  = Weight (kg) / (Height (m) \* Height (m)).

# Light Density Index (LDI)

The Light Density Index (LDI) is defined, for each zone to be treated, as the ratio of the cumulative length of illumination tip of the fibres (in cm) per cubic centimeter of the targeted zone. It is calculated as:

TI = (Total length of illumination tip of the fibre)/treatment volume

#### Where:

- > The Total length of illumination tip of the fibre is the sum of the length of each illumination tip of the fibres used during the procedure for the treated lobe or quadrant. The volume of the targeted zone is calculated precisely by the prostate MRI conducted pre-treatment.
- > An LDI equal or superior to 1.0 should be achieved for each zone to be treated.

# Baseline value

Baseline value will be defined as the last reported value until the date of treatment.

For those patients with two biopsies at baseline the following definitions of baseline values will be applied: Baseline number of positive cores

Maximum number of positive cores in the left lobe across both biopsies + maximum number of positive cores in the right lobe across both biopsies.

# Baseline maximum cancer core length

Maximum cancer core length in the left lobe across both biopsies + maximum cancer core length in the right lobe across both biopsies.

# Baseline total cancer core length

Maximum total cancer core length in the left lobe across both biopsies + maximum total cancer core length in the right lobe across both biopsies.

CLIN1601 PCM204 SAP 

# Handling of missing data and/or invalid data and outliers

#### **IIEF** questionnaire

Subscale scores with at least 1 but not more than 50% missing items will be imputed using the formula:  $S = s \times T \div t$  where s is the observed score, S is the imputed score, T is the maximum total score for the subscale and t is the maximum score possible from the completed questions. Missing subscale scores will be imputed using a multiple imputation method (Markov Chain Monte Carlo method).

# **IPSS** questionnaire

Scores with at least 1 but not more than 50% missing items will be imputed using the formula:  $S = s \times T \div t$  where s is the observed score, S is the imputed score, T is the maximum total score for the IPSS and t is the maximum score possible from the completed questions. Missing total scores will be imputed using a multiple imputation method (Markov Chain Monte Carlo method).

Other missing data, including biopsy data, will not be replaced.

A subject with missing Month 12 biopsy will be counted as failure for the primary analysis.

# Statistical plan and methods

All analysis will be carried out using contemporary versions of Stata or R.

The data collected in this study will be listed for each subject and summarized as appropriate for each treatment group as described below.

Continuous variables will be described using: number of available observations, median, first quartile (Q1), third quartile (Q3) using three significant figures.

Qualitative variables will be summarized by number of observations and percentages (%). Percentages will be rounded to two significant figures and will be based on available observations, unless otherwise specified.

## Background characteristics

# **Subject disposition**

The overall number of screen failures will be presented.

The number of subjects consented, who completed the study, who discontinued early and the reasons for early terminations will be summarized by treatment group.

The number of subjects recieving retreatment at 3 months will be presented.

# Demographic and baseline characteristics

Demographic characteristics such as age, gender, ethnic origin, height, weight and BMI will be summarized. Specific baseline disease characteristics such as time since diagnosis, TNM staging, PSA, prostate volume, type of disease (unilateral/bilateral), total number of positive cores will be summarized.

#### **Treatment modalities**

The number of fibres used, the energy applied and the light density index will be summarized for the VTP treatment group using standard descriptive statistics.

#### Efficacy analysis

All analyses will include the "efficacy population" as described above with s secondary analysis including patients undergoing retreatment at 3 months.

CLIN1601 PCM204 SAP 

# Primary efficacy analysis

The proportion of patients with no pattern 4 or 5 found in the 12 month biopsy will be reported along with a one-sided 90% confidence interval. Patients who have pattern 4 or 5 found before 12 months and who receive radical therapy will be treated as treatment failures. The treatment will be considered a success if the lower bound, rounded to 0.01, is 70% or higher. For a sample size of 44, this means that treatment will be declared a success if 35 or more patients respond.

#### Secondary efficacy analysis

## **Biopsy results**

Biopsy results at each follow-up (3, 12, 24, 36, 48 and 60) for each definition of positive biopsy will be given as cumulative frequency, along with 95% C.I., with radical therapy as a competing risk. The alternative definitions of positive biopsy are:

- 1. Presence of any pattern 4 or 5 disease (primary endpoint)
- 2. Presence of cancer of any grade
- 3. Presence of any pattern 4 or 5 disease in the treated lobe
- 4. Presence of cancer of any grade in the treated lobe

Analyses will be repeated with radical treatment counted as an event. As retreatment at 3 months is allowed, 3 month results will be treated as a binary endpoint with 95% C.I. presented in a table.

# Initiation of additional therapy

Additional prostate cancer treatment is defined as any treatment for prostate cancer other than TOOKAD® Soluble-VTP, including surgery, radiotherapy (external beam, brachytherapy, focused), high intensity focused ultrasound, cryotherapy, hormonal therapy for cancer, chemotherapy for cancer.

The time to initiation of therapy will be analyzed using Kaplan-Meier estimates, presented as a survival curve with corresponding 95% confidence intervals. Subjects who did not initiate any therapy will be censored at the time of study termination. The corresponding Kaplan-Meier curve will also be presented. As a sensitivity analysis, this analysis will be repeated excluding ablative therapies and hormonal therapy, that is, an analysis of time to radical therapy (surgery, radiotherapy). Tables and figures will be provided as appropriate.

## Safety analysis

All safety analyses will be based on the safety population. A secondary analysis will include only those patients receiving retreatment at 3 months. Results will be tabulated.

#### Adverse events

Distinctions will be made between the adverse events not related to the study treatment, related to the study treatment or related to the technical procedure of the VTP. Frequencies of AEs will be tabulated by treatment arm and the proportions of patients exhibiting each AE will be displayed. The adverse events will be classified according to MedDRA version 23.1 or higher.

The treatment-emergent adverse events (adverse events starting after the treatment) will be summarized by System Organ Class (SOC) and preferred term. In addition, the adverse events will be classified according to the NCI Common Terminology Criteria for Adverse Events which is a safety end point of the study. Tabulations will also be made for the System Organ Class, intensity, relationship, seriousness, and attribution corresponding to each AE. Separate tabulations will be made for SAEs.

CLIN1601 PCM204 SAP 

## IPSS (International Prostate Symptom Score) questionnaire

The IPSS score will be calculated as the sum of answers to questions 1 to 7. Prostate related quality of life will be derived from question 8. Descriptive summaries of change from baseline scores at each assessment visit will be provided for both Observed Cases and a multiple imputation method approaches.

# IIEF (International Index of Erectile Function) questionnaire

All items will be scored in 5 domains as follows:

- Frectile Function: sum of items 1, 2, 3, 4, 5 and 15 (score range: 1-30).
- Orgasmic Function: sum of items 9 and 10 (score range: 0-10).
- Sexual Desire: sum of items 11 and 12 (score range: 2-10).
- Intercourse Satisfaction: sum of items 6, 7 and 8 (score range: 0-15).
- Overall Satisfaction: sum of items 13 and 14 (score range: 2-10).

Descriptive summaries of the change from baseline will be provided for both Observed Cases and a multiple imputation method approaches.

In addition the erectile function score will be dichotomized as 22 or above vs. 21 and below and the proportion of cases with new onset erectile dysfunction at each timepoint (i.e. baseline score ≥22 but follow-up score < 22) will be reported. For a secondary analysis, new onset erectile dysfunction will be described as baseline score ≥22, follow-up score <22 and change from baseline of more than 2 points.

#### **Clinical laboratory evaluation**

Laboratory values will be individually listed by patient number. Values outside the laboratory reference ranges will be flagged on these individual data tables. The investigator will assess whether the values outside of the reference ranges are clinically significant or clinically non-significant. Lab abnormalities will be graded using the NCI Common Terminology Criteria for Adverse Events.

For those parameters that can be graded according to the NCI Common Terminology Criteria for Adverse Events, summaries of shift from baseline in toxicity grade to each post-baseline visit will be provided. For those parameters that cannot be graded, frequencies of patients' transitions between normal and abnormal not clinically significant (NCS) and abnormal clinically significant (CS) categories will be tabulated.

#### Vital signs

Descriptive statistics for raw and change from baseline at each planned assessment will be provided by treatment group for oral temperature, blood pressure and pulse rate using both the continuous measure and the proportion of patients outside the reference range (>38°C, >120/80 and 60 – 100, respectively) and will be presented in a table.

## Physical exam

All physical examination data and abnormalities will be listed.

## Changes from the planned analysis in study protocol

## References

The documents used to prepare this SAP include:

➤ MSKCC IRB protocol 17-070 A(2)

CLIN1601 PCM204 SAP 



Status: Completed

## **Certificate Of Completion**

Envelope Id: B33B715F962A4D0F88AC5BEDAA6ED599

Subject: Please DocuSign: PCM204\_SAP\_22DEC20.doc

Source Envelope:

Document Pages: 10 Signatures: 2 Envelope Originator: Certificate Pages: 5 Initials: 0 Suzanne Wilson

AutoNav: Enabled s.wilson-ext@stebabiotech.com IP Address: 68.83.249.159 Envelopeld Stamping: Enabled

Time Zone: (UTC+01:00) Brussels, Copenhagen, Madrid, Paris

**Record Tracking** 

Status: Original Holder: Suzanne Wilson Location: DocuSign

12/31/2020 3:59:06 PM s.wilson-ext@stebabiotech.com

**Signer Events Signature Timestamp Andrew Vickers** Sent: 12/31/2020 4:02:58 PM Andrew Victors vickersa@MSKCC.ORG Viewed: 1/4/2021 5:30:07 PM Signed: 1/4/2021 5:30:47 PM Attending

Dr. Andrew Vickers

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

723A6CE1-89A1-49B1-9E54-2AC8A75D3229

Using IP Address: 140.163.254.158

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 1/4/2021 5:30:07 PM

ID: dfc4e106-f9f0-4599-a09a-92fda77cad5c

Simon Hogan Sent: 1/4/2021 5:30:49 PM Simon Hogan s.hogan@stebabiotech.com Viewed: 1/4/2021 5:31:41 PM Signed: 1/4/2021 5:32:05 PM

EU Medical Affairs Lead STFBA Biotech

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

D37CB9E9-BA4D-47E7-A839-85580847AB82

Using IP Address: 151.226.30.116

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 10/13/2020 11:01:23 AM

ID: 1459875c-5782-40d3-8431-ea1c0b4d5a5b

| In Person Signer Events | Signature | Timestamp |
|------------------------------|-----------|-----------|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |

| Carbon Copy Events | Status | Timestamp |
|---|---|---|
| Witness Events | Signature | Timestamp |
| Notary Events | Signature | Timestamp |
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 12/31/2020 4:02:58 PM |
| Certified Delivered | Security Checked | 1/4/2021 5:31:41 PM |
| Signing Complete | Security Checked | 1/4/2021 5:32:05 PM |
| Completed | Security Checked | 1/4/2021 5:32:05 PM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Steba Biotech CFR part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

# Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

## Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

# Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us

# All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

# **How to contact Steba Biotech CFR part 11:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: g.camenen@stebabiotech.com

# To advise Steba Biotech CFR part 11 of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at g.camenen@stebabiotech.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

# To request paper copies from Steba Biotech CFR part 11

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to g.camenen@stebabiotech.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

# To withdraw your consent with Steba Biotech CFR part 11

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to g.camenen@stebabiotech.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

# Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

# Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send
  this Electronic Record and Disclosure to a location where you can print it, for future
  reference and access; and
- Until or unless you notify Steba Biotech CFR part 11 as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Steba Biotech CFR part 11 during the course of your relationship with Steba Biotech CFR part 11.